CLINICAL TRIAL: NCT03367741
Title: A Randomized Phase 2 Study of Cabozantinib in Combination With Nivolumab in Advanced, Recurrent Metastatic Endometrial Cancer
Brief Title: Cabozantinib S-malate and Nivolumab in Treating Patients With Advanced, Recurrent, or Metastatic Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-02211; NCI-2017-02211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-099; 10104 (Other: University Health Network Princess Margaret Cancer Center LAO); 10104 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Advanced Endometrial Carcinoma; Metastatic Endometrial Carcinoma; Recurrent Endometrial Carcinoma; Stage III Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8; Stage IV Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8
MeSH Terms: conditions — Endometrial Neoplasms; Carcinosarcoma | interventions — Biopsy; Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (cabozantinib s-malate, nivolumab) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15, then on day 1 beginning cycle 5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, and blood sample collection throughout the study and undergo biopsy at screening and optionally at follow up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm B (nivolumab) (Experimental): Patients receive nivolumab as in Arm A. Patients may cross-over to Arm A at the time of disease progression. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, and blood sample collection throughout the study and undergo biopsy at screening and optionally at follow up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm A (cabozantinib s-malate, nivolumab)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This randomized phase II trial studies how well cabozantinib s-malate and nivolumab work in treating patients with endometrial cancer that has come back (recurrent) or spread to other places in the body (advanced or metastatic). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib and nivolumab may work better in treating endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical anti-tumor activity of cabozantinib s-malate (XL184 ([cabozantinib]) and nivolumab based on progression free survival (PFS) in patients with advanced, recurrent or metastatic endometrial cancer previously treated with at least one line of platinum-based chemotherapy compared to patients receiving nivolumab alone.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of XL184 and nivolumab in terms of overall response rate (ORR) compared to nivolumab alone.

II. To evaluate overall survival (OS) of patients receiving XL184 and nivolumab compared to patients receiving nivolumab alone.

III. To evaluate the safety of combination treatment using XL184 and nivolumab in patients with advanced, recurrent metastatic endometrial cancer.

IV. To evaluate correlation between PD-L1 expression, CD3, CD4 and CD8 infiltrates and outcome (PFS, ORR, OS).

V. To compare PD-L1 expression, CD3, CD4 and CD8 infiltrates in the primary tumor (archival tissue) and in the tissue from baseline biopsy.

VI. To assess activity (PFS, ORR and OS) of nivolumab alone or in combination with XL184 according to microsatellite instability (MSI)/mismatched repair (MMR) status.

EXPLORATORY OBJECTIVES:

I. To assess activity (PFS, ORR and OS) of XL184 and nivolumab in patients progressed after previous exposure to anti PD-1, PD-L1 or PD-L2 agents or crossed-over from single agent nivolumab, and in patients with diagnosis of carcinosarcoma.

II. To compare microsatellite (MS) and MMR status, in the primary tumor (archival tissue) and in the tissue from baseline biopsy.

III. To assess the genomic and immune-markers landscape at baseline on tumor tissue and changes in immune landscape in peripheral blood during treatment and correlate with outcome.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28 and nivolumab intravenously (IV) over 30 minutes on days 1 and 15, then on day 1 beginning cycle 5. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), and blood sample collection throughout the study and undergo biopsy at screening and optionally at follow up.

ARM B: Patients receive nivolumab as in Arm A. Patients may cross-over to Arm A at the time of disease progression. Patients undergo CT scan, MRI, and blood sample collection throughout the study and undergo biopsy at screening and optionally at follow up.

In both arms, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30-37 days, then every 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed epithelial endometrial carcinoma; all histologies are accepted; patients with diagnosis of endometrial carcinosarcoma will be enrolled in the exploratory cohort (arm C) and will receive combination of cabozantinib and nivolumab
* Patients must have advance, recurrent or metastatic endometrial cancer
* Patients must have radiological evidence of disease progression following the most recent treatment
* Patients must have measurable disease according Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria
* Must have MS/MMR result available at time of registration; MS/MMR status is to be determined per local practice (i.e. immunohistochemistry [IHC], polymerase chain reaction [PCR], or other methods)
* Prior therapy: eligible subjects must have had at least one line of platinum-based chemotherapy; this may be adjuvant therapy or first line of cytotoxic therapy for metastatic disease; prior hormonal therapy for metastatic/recurrent disease, prior targeted therapy, and prior radiotherapy are allowed; no maximum number of previous lines of chemotherapies; concomitant chemo-radiation is not considered as previous line of systemic chemotherapy
* Availability of archival tissue for correlative analysis
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of cabozantinib and nivolumab in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 ULN (upper limit of normal), unless due to Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< 1.5 ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Serum albumin >= 28 g/L
* Lipase =< 2 ULN
* Urine protein/ creatinine ratio (UPCR) =< 1
* Prothrombin time (PT)/ international normalized ratio (INR) and partial thromboplastin time (PTT) test =< 1.3 ULN
* Patient must have disease amenable to biopsy and must agree to have one baseline biopsy
* The effects of cabozantinib and nivolumab on the developing human fetus are unknown; women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test at screening; WOCBP must agree to use adequate contraception (barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 7 months after the last dose of investigational drug; women must not be breastfeeding; women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* CROSS-OVER ELIGIBILITY CRITERIA
* Patient must provide a tumor biopsy at the time of progression on Arm B; if a patient does not have a tumor lesion amenable to biopsy or it has been unsafe for a biopsy to be performed, cross-over will not be allowed

Exclusion Criteria:

* Patients who have had chemotherapy (including investigational cytotoxic chemotherapy), biologic agents (e.g. targeted therapy or antibodies) or radiotherapy within 4 weeks prior to the first dose of study treatment
* Patients who have not recovered from adverse events attributed to prior anti-cancer therapy (i.e. have residual toxicities > grade 1, except for alopecia, neuropathy, lymphocytopenia and other non-clinically significant adverse events)
* Patients who are receiving any other investigational agents
* Patients should be excluded if they have had prior treatment with anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation; previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 is allowed and patients will be enrolled in the exploratory cohort (arm C) at the time of progression from last line of treatment (treatment with immune check point inhibitor does not have to necessary be the last line of treatment)
* Patients should be excluded if they have had prior treatment with cabozantinib; previous use of other antiangiogenic agents other than cabozantinib is allowed
* Any other active malignancy other than the endometrial cancer, that is progressing or requiring active treatment with the exception of basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because of the possible increased risk of bleeding if treatment with antiangiogenic agents is provided; patients with history of brain metastases can enroll provided the brain metastases were removed and controlled with no radiological evidence within the past 6 months
* Patients requiring concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor Xa inhibitors, antiplatelet agents (e.g. clopidogrel) or new oral anticoagulants; low-dose aspirin (=< 81 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib or nivolumab
* Patients require chronic concomitant treatment of strong CYP450 3A4 inducers (e.g. dexamethasone, phenytoin, carbamazepine, rifampicin, rifabutin, rifapentine, phenobarbital, St. John's wort) or inhibitors (e.g. ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil and conivaptan); because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list, medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment;
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment;
  * Any other signs indicative of hemorrhage within 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of XL184 (cabozantinib)
* Subject with extensive pelvic mass at risk of fistulization, or history of bowel obstruction within 3 months prior to the proposed first dose of study treatment
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * Intra-abdominal tumor/metastases invading GI mucosa
      * Active peptic ulcer disease,
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      * Malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Intra-abdominal abscess; Note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
* Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement
* Other clinically significant disorders such as:

  * Active infection requiring systemic treatment within 28 days before the first dose of study treatment
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
  * History of major surgery as follows:

    * Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
    * Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications
  * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* Known active human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS) related illness, or hepatitis B or C infection
* Administration of a live vaccine within 4 weeks prior to start of protocol therapy
* Subjects with diagnosis of immunodeficiency or who are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; the following are exceptions to this exclusion criteria: intranasal, inhaled, topical steroids, or local steroids injections (e.g. intra-articular injection); systemic corticosteroids at physiologic dose not to exceed 10 mg/day of prednisone or equivalent; steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History of autoimmune disease, such as, but not restricted to: rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematous, ankylosing spondylitis, scleroderma, or multiple sclerosis requiring treatment within the last two years; patients with vitiligo or diabetes are not excluded; replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; patients with recent history of thyroiditis; subjects with remote history (greater than 5 years) of thyroiditis are not excluded
* Psychiatric illness/social situations that would limit compliance with study requirements
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization; Note: if initial QTcF is found to be > 500 ms, two additional electrocardiogram (EKG)s separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
* Patient is not able to swallow pills
* Pregnant women are excluded from this study because XL184 and nivolumab are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with XL184 and nivolumab, breastfeeding should be discontinued if the mother is treated with XL184 and nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2026-07-23 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 1 year

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  Summary statistics, such as mean, median, counts and proportion, will be used to summarize the patients. Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon rank sum test may be substituted if necessary. 95% percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Overall survival (OS) | Up to 1 year
  Survival estimates will be computed using the Kaplan-Meier method.
Incidence of adverse events | Up to 1 year
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
PD-L1 expression, CD3, CD4 and CD8 analysis | Up to 1 year
  Correlated with outcomes (PFS, ORR, OS). The log rank test, cox model or Chi-Square test will apply to access the association between PD-L1, CD3, CD4, CD8 expression and outcome (PFS, OS, ORR) where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (34):
- United States (33):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lheureux S, Matei DE, Konstantinopoulos PA, Wang BX, Gadalla R, Block MS, Jewell A, Gaillard SL, McHale M, McCourt C, Temkin S, Girda E, Backes FJ, Werner TL, Duska L, Kehoe S, Colombo I, Wang L, Li X, Wildman R, Soleimani S, Lien S, Wright J, Pugh T, Ohashi PS, Brooks DG, Fleming GF. Translational randomized phase II trial of cabozantinib in combination with nivolumab in advanced, recurrent, or metastatic endometrial cancer. J Immunother Cancer. 2022 Mar;10(3):e004233. doi: 10.1136/jitc-2021-004233. PMID 35288469